CLINICAL TRIAL: NCT04650529
Title: G-NUH (Gyeongsang National University Hospital) Registry
Brief Title: Gyeongsang National University Hospital Registry
Acronym: GNUH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Hoon Jeong, Director, Cardiovascular Center, Gyeongsang National University Hospital
Other Study IDs: G-NUH
Record Dates: First submitted 2020-11-23; First posted 2020-12-02 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Percutaneous Coronary Intervention; Hemostatic Disorder; Blood Clot
Keywords: East Asian Paradox
MeSH Terms: conditions — Hemostatic Disorders; Thrombosis | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — After we receive patients' approval, their blood would be collected before PCI. The blood will be stored in Biobank (Gyeongsang National University Hospital).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: stent, ballooning — DES, BMS, BRS, DEB, and POBA can be used for PCI

SUMMARY:
The G-NUH registry is a two-center, real-world registry of percutaneous coronary intervention in patients with significant coronary artery disease. From January 2010, PCI-treated patients from Gyeonsang National University Hospitals (Jinju & Changwon) were enrolled in this registry.

The aim of this registry is to investigate long-term clinical outcomes and predictors of adverse outcomes after percutaneous coronary intervention from the academic hospitals.

DETAILED DESCRIPTION:
In the G-NUH registry, the investigators have collected and measured multiple hemostatic, physiologic and laboratory measurements (on-admission & 1-month) and questionnarred from PCI-treated patients. This registry will focus on the impacts of these parameters on long-term clinical outcomes from East Asian patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Significant coronary artery disease
* Treated with PCI
* Multiple hemostatic or physiologic measurements

Exclusion Criteria:

* Medically treated cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The GNUH registry is focused on clinical impact of multiple hemostatic, physiologic and laboratory measurements on CAD patients treated with PCI.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MACE | up to 10 years
  the composite of cardiovascular death, myocardial infarction or stroke

SECONDARY OUTCOMES:
Cardiovascular death | up to 10 years
  Mortality related with cardiovascular events
Myocardial infarction | up to 10 years
  Fatal & non-fatal myocardial infarction
Stroke | up to 10 years
  Ischemic & hemorrhagic stroke
Revascularization | up to 10 years
  target-lesion, target-vessel vs. nontarget-vessel
Major bleeding | up to 10 years
  BARC type 3-5
Stent thrombosis | up to 10 years
  Thrombotic events in & near to stent
ISR | up to 10 years
  in-stent restenosis

OTHER OUTCOMES:
Incidence of MACE according to platelet function | up to 10 years
  VerifyNow assay
Incidence of MACE according to global hemostasis assay | up to 10 years
  thromboelastography (TEG: R, alpha angle, MA and LY30)
Incidence of MACE according to hemostatic biomarkers | up to 10 years
  hs-CRP, fibrinogen, D-dimer, NT-proBNP, lipid battery
Incidence of MACE according to cardiac contractility | up to 10 years
  Echocardiography: LV EF, E/A, TR Vmax, LAVI
Incidence of MACE according to physiologic index | up to 10 years
  fractional flow reserve (FFR), coronary flow reserve (CFR) and the index of microvascular resistance (IMR)
Incidence of MACE according to 1-month bleeding & dyspnea episodes | up to 10 years
  Qestionnarres for bleeding, dyspnea, side effects

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Jeong, MD, PhD, Study Director — Changwon Gyeongsang National University Hospital
Locations (2):
- South Korea (2):
  - Changwon Gyeongsang National University Hospital, Changwon, Gyeongsangnam-do
  - Gyeonsang National University Hospital, Jinju, Gyeonsangnam-do

IPD SHARING:
Plan to Share IPD: Undecided
This registry would be shared with other researchers in terms of whole collected data.

REFERENCES:
- [Result] Bae JS, Ahn JH, Jang JY, Cho SY, Kang MG, Kim KH, Park HW, Koh JS, Park Y, Hwang SJ, Kwak CH, Hwang JY, Tantry US, Gurbel PA, Jeong YH. The Impact of platelet-fibrin clot strength on occurrence and clinical outcomes of peripheral artery disease in patients with significant coronary artery disease. J Thromb Thrombolysis. 2020 Nov;50(4):969-981. doi: 10.1007/s11239-020-02103-w. PMID 32279217
- [Derived] Cho JH, Ahn JH, Kang MG, Bae JS, Koh JS, Jung MK, Kim SW, Gorog DA, Tantry US, Gurbel PA, Kim W, Hwang JY, Jeong YH. Residual Cardiovascular Biomarkers After Medical Therapy and Their Prognostic Implications Following Percutaneous Coronary Intervention. JACC Adv. 2026 Jan 2;5(2):102498. doi: 10.1016/j.jacadv.2025.102498. Online ahead of print. PMID 41483545
- [Derived] Omar M, Kang MG, Jung MK, Ahn JH, Koh JS, Guevarra PI, Kim SW, Tantry US, Gurbel PA, Hwang JY, Jeong YH. Association and Prognostic Implications of "No-Reflow Phenomenon" and Hypercoagulability in Patients With ST-Segment Elevation Myocardial Infarction. JACC Asia. 2025 Nov;5(11):1487-1501. doi: 10.1016/j.jacasi.2025.07.015. Epub 2025 Sep 5. PMID 40910963
- [Derived] Cho S, Jung M, Ahn JH, Kang MG, Bae JS, Koh JS, Hwang SJ, Kim HS, Kim SW, Hwang JY, Jeong YH. Diabetic Status and Thrombogenicity: Association and Prognostic Implications After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2025 Mar 24;18(6):720-733. doi: 10.1016/j.jcin.2024.12.002. PMID 40139850
- [Derived] Lee SY, Cho JY, Gorog DA, Angiolillo DJ, Yun KH, Ahn JH, Koh JS, Park Y, Hwang SJ, Hwang JY, Kim JW, Jang Y, Jeong YH. Inflammation and platelet reactivity during adjunctive colchicine versus aspirin in patients with acute coronary syndrome treated with potent P2Y12 inhibitor. Front Med (Lausanne). 2024 Apr 19;11:1349577. doi: 10.3389/fmed.2024.1349577. eCollection 2024. PMID 38841588
- [Derived] Lee SH, Kim HK, Ahn JH, Kang MG, Kim KH, Bae JS, Cho SY, Koh JS, Park Y, Hwang SJ, Gorog DA, Tantry US, Bliden KP, Gurbel PA, Hwang JY, Jeong YH. Prognostic impact of hypercoagulability and impaired fibrinolysis in acute myocardial infarction. Eur Heart J. 2023 May 14;44(19):1718-1728. doi: 10.1093/eurheartj/ehad088. PMID 36857519
- [Derived] Ahn JH, Tantry US, Kang MG, Park HW, Koh JS, Bae JS, Cho SY, Kim KH, Jang JY, Park JR, Park Y, Hwang SJ, Kwak CH, Hwang JY, Gurbel PA, Jeong YH. Residual Inflammatory Risk and its Association With Events in East Asian Patients After Coronary Intervention. JACC Asia. 2022 Apr 12;2(3):323-337. doi: 10.1016/j.jacasi.2021.11.014. eCollection 2022 Jun. PMID 36338415
- See also: Analysis from the G-NUH registry — https://link.springer.com/article/10.1007/s11239-020-02103-w